CLINICAL TRIAL: NCT07151924
Title: Eating Disturbances in Patients With Type 1 Diabetes Initiating Closed-loop Insulin Therapy: Prevalence and Influence on Glycemic Control
Brief Title: Eating Disturbances in Patients With Type 1 Diabetes Initiating Insulin Therapy
Acronym: CALI-BF
Status: Active, not recruiting | Type: Observational
Sponsor: University Hospital, Toulouse (Other)
Responsible Party: Sponsor
Other Study IDs: RC31/24/0571; ID-RCB (Other: 2025-A01127-42)
Record Dates: First submitted 2025-07-18; First posted 2025-09-03 (Actual); Last update posted 2025-09-24 (Actual); Status verified 2025-09

CONDITIONS: Diabete Type 1
Keywords: diabete type 1; eating disorders; eating; insulin; insulin therapy
MeSH Terms: conditions — Feeding and Eating Disorders; Insulin Resistance

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 6 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients with type 1 diabete: Patients with type 1 diabete with closed-loop therapy
  Interventions: Other: Questionnaires answers; Other: Biological assessment

INTERVENTIONS:
Other: Questionnaires answers — Patients will be asked to complete the MScoff and QACD questionnaires during interviews with the dietitian at baseline, 3 months and 6 months.
Other: Biological assessment — Collection of HbA1c level and continuous glucose monitoring data

SUMMARY:
The prevalence of eating disorders is particularly high among people with type 1 diabetes (T1D). These abnormalities, such as "diabulimia," are frequently responsible for poor insulin therapy management and, consequently, chronic glycemic imbalance, exposing them to an increased risk of complications. Their detection and management unfortunately remain insufficient in current practice.

However, to date, no study has addressed the question of the prevalence and impact of eating disorders in this context. Our research hypotheses are therefore as follows:

1. The existence of an eating disorder is likely frequently overlooked and, therefore, not taken into account in patients with T1D initiating semi-automated insulin therapy with BF.
2. The existence of an eating disorder could impair the performance of the BF device in terms of improving glycemic control in patients with T1D initiating this treatment method.

Patients clinical characteristics, glycemic monitoring parameters ad questionnaires answers will be recorded. The prevalence of eating disorders will be calculated, and the association between the presence of these abnormalities and baseline clinical characteristics and glycemic control parameters will be analyzed.

DETAILED DESCRIPTION:
The prevalence of eating disorders (EDs) and problematic eating behaviors (PEBs) is particularly high among people with type 1 diabetes (T1D), affecting 20 to 50% of women and 5 to 25% of men among young patients. These abnormalities, such as "diabulimia," are frequently responsible for poor insulin therapy management and, consequently, chronic glycemic imbalance, exposing them to an increased risk of complications. Their detection and management unfortunately remain insufficient in current practice.

The treatment of T1D is currently undergoing a veritable technological revolution linked to the arrival of the first semi-automated insulin therapy devices (or closed loop, LF). The use of these devices most often makes it possible to achieve recommended glycemic control targets (HbA1c, continuous glucose monitoring [CGM] data), reduce glycemic variability, and avoid hypoglycemia. Insulin administration is based on the data transmitted: food intake and quantity of carbohydrates consumed. The role of dietitians is therefore crucial in the therapeutic education of patients and the care pathway imposed by the initiation of this new treatment method. It is likely that many patients initiating automated insulin therapy with BF present an eating disorder or CAP that may interfere with the management of the device.

However, to date, no study has addressed the question of the prevalence and impact of eating disorders and CAP in this context. In the absence of available data, national and international recommendation texts dedicated to insulin therapy with BF do not specify appropriate conduct for patients presenting with these eating disorders. Our research hypotheses are therefore as follows:

1. The existence of an eating disorder (ED and/or CAP) is likely frequently overlooked and, therefore, not taken into account in patients with T1D initiating semi-automated insulin therapy with BF.
2. The existence of an eating disorder (ED and/or CAP) could impair the performance of the BF device in terms of improving glycemic control in patients with T1D initiating this treatment method.

Patients clinical characteristics and glycemic monitoring parameters (HbA1c and CGM data), available as part of routine care, will be recorded in an electronic case report (REDCap software). The mSCOFF and QACD questionnaires will be administered during the dietary interview preceding BF device implantation, and responses will be collected. The prevalence of eating disorders will be calculated, and the association between the presence of these abnormalities and baseline clinical characteristics and glycemic control parameters will be analyzed.

The care pathway established for initiating BF treatment requires a follow-up medical consultation at 3 months, followed by a consultation at 6 months. As part of the study, visits at 3 months (12 ± 2 weeks) and 6 months (24 ± 4 weeks) will be scheduled and will include an interview with a dietitian, to collect glycemic control parameters (at 3 and 6 months), measure body weight (at 3 and 6 months), and repeat the mSCOFF and QACD questionnaires (at 6 months). Data on the evolution of glycemic control and variability parameters, weight and mSCOFF and QACD scores will be analyzed in the overall study population, then according to the existence or not of disturbances in eating behavior at inclusion.

ELIGIBILITY:
Inclusion Criteria:

* Patient diagnosed with type 1 diabetes.
* Patient with a CGM device for more than 3 months with > 80% of data captured in the last month.
* Indication for the implementation of a BF device as part of routine care, in the Diabetology, Metabolic Diseases and Nutrition Department of the Toulouse University Hospital (initiating center).

Exclusion Criteria:

* Pregnant or breastfeeding women, or those planning to become pregnant within 6 months of inclusion.
* History of obesity surgery or a preparatory program for obesity surgery planned during the study period.
* Pharmacological treatment likely to significantly influence food intake and body weight, whether ongoing or discontinued within the last 3 months (e.g., GLP-1R agonist): Liraglutide (Victoza®, Saxenda®), Semaglutide (Ozempic®, Wegovy®), Dulaglutide (Trulicity®), Tirzepatde (Mounjaro®), Orlistat (Xenical®)
* Eating disorder requiring specific treatment in the previous 12 months.
* Refusal or inability to consent to participate.
* Persons under legal protection (guardianship, curatorship, or court-ordered protection).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients with type 1 diabetes for whom closed-loop insulin therapy has been recommended
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2025-09-04 (Actual); Primary Completion 2027-02-28 (Estimated); Study Completion 2027-02-28 (Estimated)

PRIMARY OUTCOMES:
Prevalence of eating disorders | 6 months after the inclusion
  The primary outcome measure for establishing the prevalence of eating disorders is a composite outcome measure based on determining the existence of eating disorders [ED] by analyzing responses to the mSCOFF questionnaire (score ≥ 2) and/or problematic eating behaviors [PEB] by analyzing responses to the QACD questionnaire (score ≥ 20).

SECONDARY OUTCOMES:
Prevalence of eating disorders (EDs) | 6 months after the inclusion
  Prevalence of EDs (mSCOFF score ≥ 2 and QACD ≥ 20)
Clinical characteristics at inclusion | 6 months after the inclusion
  Measurement of clinical characteristics at inclusion: age
Clinical characteristics at inclusion | 6 months after the inclusion
  Measurement of clinical characteristics at inclusion: sex
Clinical characteristics at inclusion | 6 months after the inclusion
  Measurement of clinical characteristics at inclusion: weight in kg and height in cm which will be combined to calculate the BMI (kg/m²)
Clinical characteristics at inclusion | 6 months after the inclusion
  Measurement of clinical characteristics at inclusion: medical history
Clinical characteristics at inclusion | 6 months after the inclusion
  Measurement of clinical characteristics at inclusion: treatments
Description of glycemic control at inclusion | 6 months after the inclusion
  Measurement of basic glycemic control : Hba1c average
Description of variability indicators at inclusion | 6 months after the inclusion
  Measurement of basic glycemic variability parameters : continuous glucose measurement data
Evolution of biological parameters of glycemic variability between the inclusion visit and the follow-up visits | 6 months after the inclusion
  Measurement of the variation in blood glycemic variability (continuous glucose measurement data) parameters between the inclusion visit and the different follow-up visits (3 months and 6 months)
Evolution of biological control parameters variability between the inclusion visit and the follow-up visits | 6 months after the inclusion
  Measurement of the variation in blood control parameters variability (HbA1c) between the inclusion visit and the different follow-up visits (3 months and 6 months)
Evolution of BMI between inclusion and follow-up visits | 6 months after the inclusion
  Change in BMI between the baseline visit and the 3-month and 6-month follow-up visits
Evolution of body weight between inclusion and follow-up visits | 6 months after the inclusion
  Change in body weight between the baseline visit and the 3-month and 6-month follow-up visits
Change in questionnaires scores between baseline and follow-up | 6 months after the inclusion
  Change in mSCOFF (Sick, control, one stone, fat, food) scores between the baseline visit and the 6-month follow-up visit
Change in questionnaires scores between baseline and follow-up | 6 months after the inclusion
  Change in QACD (questionnaires of attitudes and behaviors related to diabetes management) scores between the baseline visit and the 6-month follow-up visit

CONTACTS AND LOCATIONS:
Locations (1):
- Diabetology, Metabolic Diseases and Nutrition Department Rangueil Hospital, Toulouse University Hospital 1 avenue du Pr Jean Poulhès, Toulouse, France

IPD SHARING:
Plan to Share IPD: No